CLINICAL TRIAL: NCT06301906
Title: Gut Microbiota and Bile Acids Mediate the Clinical Benefits of Red Yeast Rice for Primary Prevention of Hypercholesterolemia: A Pilot Observational Study
Brief Title: Red Yeast Rice for Primary Prevention of Hypercholesterolemia
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301060A3
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — BID protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: LipoCol Forte Capsule 600mg bid

INTERVENTIONS:
Drug: LipoCol Forte Capsule 600mg bid — LipoCol Forte Capsule 600mg bid for 12 months

SUMMARY:
This two-year observational study will be conducted at the outpatient clinic of the Department of Traditional Chinese Medicine of Taoyuan Chang Gung Hospital from February 26, 2024 to December 31, 2025. This study will enroll 35~55 year-old male patients who are expected to take LipoCol Forte Capsules for primary prevention of hypercholesterolemia. The investigators will collect the TCM constitution questionnaires from patients before taking LipoCol Forte Capsules and every three months after taking the medicine. At the same time, blood will be drawn to detect glycated hemoglobin, fasting blood sugar, insulin, lipids profile, liver and kidney function, creatine kinase, predictive parameters of atherosclerotic cardiovascular disease, and plasma bile acids, etc. Fecal samples will also be collected to analyze the intestinal microbiota and fecal bile acid composition. This study will evaluate the efficacy, durability and safety of LipoCol Forte capsules in the primary prevention of hypercholesterolemia in patients with different constitutions, as well as whether it can reduce the risk of cardiovascular disease, and its influence on bile acid metabolism and intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35~55 years old, LDL-C≥130mg/dl or patients with diabetes or chronic kidney disease with LDL-C ≥ 100mg/dl, expected to receive LipoCol Forte Capsule 600mg bid

Exclusion Criteria:

1. Have received anti-hyperlipidemic drugs or red yeast rice treatment within the past month;
2. Female;
3. Have experienced rhabdomyolysis or abnormal liver function ALT >72 U/L due to taking red yeast rice;
4. Bleeding diseases, such as abnormal platelets, abnormal coagulation factors, or gastrointestinal tract infection within one month
5. Liver insufficiency ALT >72 U/L or renal insufficiency eGFR < 30 mL/min/1.73 m2;
6. Have ever had coronary heart disease, myocardial infarction or cerebrovascular disease;
7. Stressful situations, including hospitalization or surgery within the past or next month, and cancer still being treated;
8. Uncontrolled hypertension (blood pressure ≥160/100 mmHg);
9. Use antibiotics, probiotics or weight-loss drugs for more than 3 consecutive days within 3 months before inclusion in the study;
10. Drug abuse or poor compliance;
11. Use of traditional Chinese medicine in the past month

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators will collect the TCM constitution questionnaires from patients before taking LipoCol Forte Capsules and every three months after taking the medicine. At the same time, blood will be drawn to detect glycated hemoglobin, fasting blood sugar, insulin, lipids profile, liver and kidney function, creatine kinase, predictive parameters of atherosclerotic cardiovascular disease, and plasma bile acids, etc. Fecal samples will also be collected to analyze the intestinal microbiota and fecal bile acid composition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Low Density Lipoprotein-Cholesterol (LDL-C) | before treatment, and 3, 6, 9, 12 months after treatments
  This study will evaluate the efficacy and durability of LipoCol Forte capsules in the primary prevention of hypercholesterolemia.

SECONDARY OUTCOMES:
10-Year ASCVD Risk | before treatment, and 3, 6, 9, 12 months after treatments
  use ASCVD risk estimator to calculate the 10-Year ASCVD Risk after LipoCol Forte capsules treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan branch of Chang Gung Memorial Hospital, Taoyuan District, Taiwan